CLINICAL TRIAL: NCT00314236
Title: A Randomized, Comparative Multicenter Clinical Trial Evaluating BST-CarGel™ and Microfracture in Repair of Focal Articular Cartilage Lesions on the Femoral Condyle
Brief Title: Trial Comparing BST-CarGel and Microfracture in Repair of Articular Cartilage Lesions in the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piramal Healthcare Canada Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CG-CIP01-P
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Knee Injuries
Keywords: Cartilage repair; Cartilage; Knee; Knee Pain; Microfracture; arthroscopy; bone marrow stimulation; Chondrogenesis; Scaffold; Chitosan; A02.165.165; A10.165.382.332; G07.574.500.325.377.625.180; A10.165.382.400; Articular Cartilage Repair
MeSH Terms: conditions — Knee Injuries; Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microfracture with BST-CarGel (Experimental): BST-CarGel applied to a Microfractured lesion in repair of focal articular cartilage lesions on the femoral condyle
  Interventions: Device: BST-CarGel with Microfracture
- Microfracture without BST-CarGel (Active Comparator): Microfractured lesion in repair of focal articular cartilage lesions on the femoral condyle
  Interventions: Procedure: Microfracture without BST-CarGel

INTERVENTIONS:
Device: BST-CarGel with Microfracture — Microfracture performed with BST-CarGel added to the treated defect
  Arms: Microfracture with BST-CarGel
Procedure: Microfracture without BST-CarGel — Microfracture performed without BST-CarGel added to the treated defect.
  Arms: Microfracture without BST-CarGel

SUMMARY:
This study will investigate whether the treatment of damaged cartilage in the knee with BST-CarGel will increase the amount and quality of cartilage repair tissue when compared with microfracture alone. Furthermore, the effect of BST-CarGel in decreasing cartilage related pain and improving cartilage-related function in the knee will be assessed.

DETAILED DESCRIPTION:
Cartilage repair currently remains a problematic orthopedic concern with no effective solution. The development of new surgical techniques or therapies is critical in meeting this medical need.

This Canadian trial will be a pivotal protocol study, conducted as a randomized, controlled trial. A total of 80 subjects, 40 subjects in each of the two groups (BST-CarGel applied to a microfractured lesion or microfracture alone), will be enrolled in this study. The subjects and investigative medical staff will not be blinded to treatment due to the difference in surgical incision size. However, although the treatment will not be blinded, the primary effectiveness assessment will be blinded. The primary endpoint of this study will be cartilage repair at 12 months proved by demonstrating that BST-CarGel treatment effectively fills cartilage lesions with high quality cartilaginous tissue. The secondary endpoints will be pain, stiffness and function while other tertiary endpoints will include safety, quality-of-life (QOL), as well as macroscopic characterizations of tissue repair. The primary measure of this study will occur at 12 months, when imaging of repair tissue using magnetic resonance (MR) and associated analyses will compare tissue volume, quality and other anatomical variables. Radiographic evaluations will be blinded. Volunteer biopsies at 13 months may be obtained. Pain, stiffness, function and QOL will be assessed prior to treatment, and at 3, 6 and 12 months following treatment using self-administered validated scores (WOMAC and SF-36). In addition, subject safety will be assessed through a record of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age
* Focal articular cartilage lesion on the medial femoral condyle
* Grade 3 or 4 acute (traumatic) or chronic (degenerative) lesion
* Stable knee

Exclusion Criteria:

* Multiple lesions or kissing lesions
* Clinically relevant compartment malalignment (> 5 degrees)
* Undergone ligament treatments in the affected knee within 2 years prior to trial
* Inflammatory arthropathy, such as rheumatoid arthritis, systemic lupus, or active gout
* Previous surgical cartilage treatments in the affected knee in the last 12 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2005-12; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Stanish, MD, Principal Investigator — Orthopaedic and Sport Medicine - Dalhousie University
Locations (18):
- Canada (11):
  - Sports Medicine Centre - University of Calgary, Calgary, Alberta
  - New West Sports Medicine, New Westminster, British Columbia
  - Hospital at UBC, Vancouver, British Columbia
  - Pan Am Clinic, Winnipeg, Manitoba
  - Orthopaedic and Sport Medicine Clinic of Nova Scotia, Halifax, Nova Scotia
  - Entralogix Clinical Group Inc., Newmarket, Ontario
  - Sports Medicine Clinic - Carleton University, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Div. of Orthopaedic Surgery, Toronto, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hospital Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire de Quebec et Hôpital Valcartier, Québec, Quebec
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
- Spain (5):
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Universitario Gregorio Maraňón, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - FREMAP Centro de Prevención y Rehabilitación, Majadahonda, Madrid
  - Hospital Begona de Gijon, Gijón, Principality of Asturias

REFERENCES:
- [Background] Hoemann CD, Hurtig M, Rossomacha E, Sun J, Chevrier A, Shive MS, Buschmann MD. Chitosan-glycerol phosphate/blood implants improve hyaline cartilage repair in ovine microfracture defects. J Bone Joint Surg Am. 2005 Dec;87(12):2671-2686. doi: 10.2106/JBJS.D.02536. PMID 16322617
- [Background] Chevrier A, Hoemann CD, Sun J, Buschmann MD. Chitosan-glycerol phosphate/blood implants increase cell recruitment, transient vascularization and subchondral bone remodeling in drilled cartilage defects. Osteoarthritis Cartilage. 2007 Mar;15(3):316-27. doi: 10.1016/j.joca.2006.08.007. Epub 2006 Sep 26. PMID 17008111
- [Background] Hoemann CD, Sun J, McKee MD, Chevrier A, Rossomacha E, Rivard GE, Hurtig M, Buschmann MD. Chitosan-glycerol phosphate/blood implants elicit hyaline cartilage repair integrated with porous subchondral bone in microdrilled rabbit defects. Osteoarthritis Cartilage. 2007 Jan;15(1):78-89. doi: 10.1016/j.joca.2006.06.015. Epub 2006 Aug 8. PMID 16895758
- [Result] Stanish WD, McCormack R, Forriol F, Mohtadi N, Pelet S, Desnoyers J, Restrepo A, Shive MS. Novel scaffold-based BST-CarGel treatment results in superior cartilage repair compared with microfracture in a randomized controlled trial. J Bone Joint Surg Am. 2013 Sep 18;95(18):1640-50. doi: 10.2106/JBJS.L.01345. PMID 24048551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from May 04, 2006 to January 2009 from orthopaedic surgeon referrals across 24 centers across Canada, Europe, and South Korea.
Pre-assignment Details: Subjects were stratified by site and lesion type (acute/chronic) to address possible repair differences. Final eligibility and lesion type were determined during diagnostic arthroscopy at treatment visit, subjects were randomized to BST-CarGel or MFX treatment using a computer-generated randomization schedule to ensure a 1:1 ratio within each site.
Groups:
- Experimental: BST-CarGel applied to a Microfractured lesion
- Control: Microfracture alone
Period: Overall Study
Arm/Group | Experimental | Control
Started | 41 | 39
Completed | 41 | 37
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 39 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (9.6) | 37.2 (10.6) | 36.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 23 | 25 | 48
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 32 | 65
  Spain | 7 | 6 | 13
  Korea, Republic of | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Degree of Filling of the Lesion by Repair Tissue at 12 Months Through MRI.
Description: Evaluate the efficacy of BST-CarGel® applied to a microfractured lesion as compared to microfracture alone on the degree of lesion filling of the study knee in subjects with symptomatic pain associated with cartilage damage using MRI scans. The MR images will be acquired using high resolution 3D cartilage imaging sequences, so-called cartilage morphology sequences.
Time Frame: 12 months
Population: Sample size for degree of lesion filling was calculated using a standard t test, with an anticipated relevant difference of 15% between treatments and a common SD of 15. Under these assumptions, the sample size per group was calculated to be 23 subjects (or 46 subjects in total)
Measure: Least Squares Mean (Standard Error); unit: Percentage of lesion fill
Arm/Group | Experimental | Control
Number analyzed (Participants) | 41 | 37
Percentage of lesion fill | 92.81 (1.98) | 85.22 (2.08)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority or Other; p = 0.011, ANCOVA

2. Primary Outcome: Repair Cartilage T2 Relaxation Time
Description: Evaluate the efficacy of BST-CarGel® applied to a microfractured lesion as compared to microfracture alone on the repair tissue quality of the study knee in subjects with symptomatic pain associated with cartilage damage using MRI T2 mapping. T2 maps are created by calculating the T2 relaxation times for repair tissue and cartilage plates for every voxel (picture element of a MRI scan containing the average signal information of a specific spatial location of the imaged body).
Time Frame: 12 months
Population: Sample size for repair tissue quality was calculated, using a standard t test, with an anticipated relevant difference of 15% between treatments and a common SD of 10. Under these assumptions, the sample size per group was calculated to be 11 subjects (or 22 subjects in total)
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Experimental | Control
Number analyzed (Participants) | 41 | 37
milliseconds | 70.46 (4.49) | 85.04 (4.89)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority or Other; p = 0.033, ANCOVA

3. Secondary Outcome: Change From Baseline for Knee-related Pain, Stiffness and Function at 12 Months (WOMAC Parts A, B, C)
Description: The three sub-scales: 1) Pain, 2.) stiffness and 3.) function scores ranged from 0-10. Pain had 5 items and stiffness had 2 items, and function had 17 items. The total score for pain ranged from 0 no pain to 50 worst pain. The total score for stiffness ranged from 0 no stiffness to 20 worst stiffness. The total score for function raged from 0 no function to 170 worst function.
Time Frame: 12 months
Population: Secondary efficacy was evaluated based on pain, stiffness, and function, as well as the macroscopic nature of the cartilage repair. Measurements of pain, stiffness, and function were made at 3, 6, and 12 months post-treatment using the WOMAC questionnaire and SF-36v2. WORMS scoring was conducted on 12-month post-treatment MRI scans.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 41 | 37
Units on a scale
  Pain | -16.16 (1.16) | -16.91 (1.21)
  Stiffness | -5.97 (0.68) | -6.56 (0.71)
  Function | -55.96 (4.24) | -60.59 (4.41)

4. Secondary Outcome: Frequency of Adverse Events Between Study Groups
Time Frame: 12 months
Population: AEs will be coded and tabulated separately by system organ class (SOC) and individual preferred terms (PTs). The number and percentage of subjects who experienced AEs will be summarized in decreasing frequency by using the medical dictionary for regulatory activities (MedDRA) dictionary.
Measure: Number; unit: Percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 41 | 39
Percentage of participants | 97.6 | 92.3

ADVERSE EVENTS:
Time Frame: AEs were reported through out the study from signed Informed Consent up to 12 months post-treatment.
Description: Only subjects randomized to BST-CarGel® treatment were exposed to the investigational device.
Arm/Group | Experimental | Control
Serious Adverse Events (participants affected / at risk) | 5/41 | 1/39
Other Adverse Events (participants affected / at risk) | 40/41 | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Experimental (N=41) | Control (N=39)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/1 (2) | 0 (0) — Subject experienced pulmonary embolism. Drug therapy administered at onset, and subject recovered. All SAEs, onset of pulmonary emboli secondary to DVT and pleurisy post-treatment, considered related to the procedure and possibly related to device.
deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) — Deep vein thrombosis,classified - severe. Drug therapy administered at onset, and subject recovered.All SAEs, onset of pulmonary emboli secondary to DVT and pleurisy, post-treatment, considered related to the procedure and possibly related to device.
pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pleurisy associated to pulmonary embolism. Severe, sequelae of main SAE. Pleurisy not treated w/medication, subject recovered. All SAEs, onset of pulmonary emboli secondary to DVT and pleurisy, considered related to procedure and possibly to device.
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Subject experienced wheezing of moderate severity. Drug therapy administered at the onset of the SAE, and the subject recovered. The SAE, onset at same day post-treatment, was considered to be related to the procedure but not related to the device.
chest pain (General disorders) | 0 (0) | 1 (1) — Subject experienced chest pain of moderate severity. Drug therapy was administered at the onset of the SAE, and the subject recovered. The SAE, onset at Day 346 post-treatment, was considered to be unrelated to the procedure.
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject experienced diarrhea;classified as severe. Drug therapy was administered at the onset of the SAE, and the subject recovered. The SAE, onset at Day 151 post-treatment, was considered to be unrelated to the procedure and the device.
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject experienced joint stiffness; classified as severe. Drug therapy was administered at the onset, and subject recovered with sequelae. The SAE, onset at Day 34 post-treatment, considered to be related to procedure but not related to the device.
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject experienced joint ankylosis; classified as severe. Drug therapy was administered at onset, and subject recovered with sequelae. The SAE, onset at Day 93 post-treatment, considered possibly related to procedure but not related to the device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=41) | Control (N=39)
arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 25
joint effusion (Musculoskeletal and connective tissue disorders) | 6 | 3
joint stiffness (Musculoskeletal and connective tissue disorders) | 5 | 4
joint swelling (Musculoskeletal and connective tissue disorders) | 5 | 2
back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 1
joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
muscular spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 | 0
muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
procedural pain (Injury, poisoning and procedural complications) | 13 | 12
post-procedural nausea (Injury, poisoning and procedural complications) | 5 | 2
burns second degree (Injury, poisoning and procedural complications) | 0 | 1
epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
fall (Injury, poisoning and procedural complications) | 0 | 1
frostbite (Injury, poisoning and procedural complications) | 1 | 0
hand fracture (Injury, poisoning and procedural complications) | 0 | 1
incision site complication (Injury, poisoning and procedural complications) | 0 | 1
joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
joint injury (Injury, poisoning and procedural complications) | 1 | 0
joint sprain (Injury, poisoning and procedural complications) | 0 | 1
limb injury (Injury, poisoning and procedural complications) | 0 | 1
post-procedural edema (Injury, poisoning and procedural complications) | 1 | 0
road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
seroma (Injury, poisoning and procedural complications) | 1 | 0
headache (Nervous system disorders) | 5 | 5
dizziness (Nervous system disorders) | 3 | 2
tremor (Nervous system disorders) | 1 | 1
balance disorder (Nervous system disorders) | 1 | 0
burning sensation (Nervous system disorders) | 1 | 0
carpal tunnel syndrome (Nervous system disorders) | 1 | 0
complex regional pain syndrome (Nervous system disorders) | 0 | 1
convulsion (Nervous system disorders) | 1 | 0
disturbance in attention (Nervous system disorders) | 0 | 1
hyperesthesia (Nervous system disorders) | 1 | 0
loss of consciousness (Nervous system disorders) | 1 | 0
syncope vasovagal (Nervous system disorders) | 1 | 0
chills (General disorders) | 3 | 2
pyrexia (General disorders) | 4 | 1
influenza-like illness (General disorders) | 2 | 1
edema peripheral (General disorders) | 2 | 1
adverse drug reaction (General disorders) | 1 | 1
chest pain (General disorders) | 0 | 1
discomfort (General disorders) | 0 | 1
drug intolerance (General disorders) | 0 | 1
feeling hot (General disorders) | 0 | 1
feeling of relaxation (General disorders) | 0 | 1
injection site bruising (General disorders) | 1 | 0
injection site pain (General disorders) | 0 | 1
malaise (General disorders) | 1 | 0
pain (General disorders) | 1 | 0
nasopharyngitis (Infections and infestations) | 1 | 5
sinusitis (Infections and infestations) | 0 | 3
upper respiratory tract infection (Infections and infestations) | 1 | 2
bronchitis (Infections and infestations) | 1 | 1
infected insect bite (Infections and infestations) | 2 | 0
clostridium colitis (Infections and infestations) | 1 | 0
escherichia infection (Infections and infestations) | 1 | 0
gastroenteritis viral (Infections and infestations) | 0 | 1
gingival infection (Infections and infestations) | 1 | 0
herpes zoster (Infections and infestations) | 0 | 1
influenza (Infections and infestations) | 1 | 0
laryngitis (Infections and infestations) | 0 | 1
onychomycosis (Infections and infestations) | 1 | 0
pharyngitis (Infections and infestations) | 1 | 0
skin infection (Infections and infestations) | 1 | 0
stitch abscess (Infections and infestations) | 1 | 0
tinea pedis (Infections and infestations) | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 1
nausea (Gastrointestinal disorders) | 7 | 0
vomiting (Gastrointestinal disorders) | 5 | 0
diarrhea (Gastrointestinal disorders) | 4 | 0
constipation (Gastrointestinal disorders) | 2 | 0
abdominal pain lower (Gastrointestinal disorders) | 1 | 0
abdominal pain upper (Gastrointestinal disorders) | 1 | 0
crohn's disease (Gastrointestinal disorders) | 1 | 0
dyspepsia (Gastrointestinal disorders) | 1 | 0
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
pruritis (Skin and subcutaneous tissue disorders) | 3 | 0
acne (Skin and subcutaneous tissue disorders) | 0 | 1
eczema (Skin and subcutaneous tissue disorders) | 0 | 1
excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
keloid scar (Skin and subcutaneous tissue disorders) | 1 | 0
pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 1
rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
hypertension (Vascular disorders) | 1 | 1
circulatory depression (Vascular disorders) | 0 | 1
deep vein thrombosis (Vascular disorders) | 1 | 0
hypotension (Vascular disorders) | 0 | 1
peripheral coldness (Vascular disorders) | 0 | 1
thrombophlebitis (Vascular disorders) | 1 | 0
blood pressure decreased (Vascular disorders) | 1 | 0
blood pressure increased (Vascular disorders) | 1 | 0
body temperature increased (Vascular disorders) | 1 | 0
weight increased (Vascular disorders) | 0 | 1
anemia (Blood and lymphatic system disorders) | 2 | 1
anxiety (Psychiatric disorders) | 1 | 0
hallucination (Psychiatric disorders) | 1 | 0
dysuria (Renal and urinary disorders) | 0 | 1
polyuria (Renal and urinary disorders) | 1 | 0
vertigo (Ear and labyrinth disorders) | 0 | 1
drug hypersensitivity (Immune system disorders) | 0 | 1
podagra (Metabolism and nutrition disorders) | 1 | 0
uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
cervical dysplasia (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the Institution/PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is > 60 days but ≤ 90 days from time submitted to sponsor for review. Sponsor can require changes to communication. Control over publication/presentation shall be extended for maximum of 2 years after termination of Trial, after which Institution/PI shall be free to publish/present without restraint.